CLINICAL TRIAL: NCT05653583
Title: A Feasibility Study of Peripheral Nerve Stimulation Therapy for Atrial Fibrillation
Brief Title: Peripheral Nerve Stimulation Therapy for Atrial Fibrillation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cala Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: AFIB-01
Record Dates: First submitted 2022-11-30; First posted 2022-12-16 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Ear Protective Devices

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- Wrist Device (Active Comparator): Twice daily stimulation sessions during the 4-week treatment period
  Interventions: Device: Wrist Device
- Ear Device (Active Comparator): Twice daily stimulation sessions during the 4-week treatment period
  Interventions: Device: Ear Device
- Sham Device (Sham Comparator): Twice daily "stimulation" sessions during the 4-week treatment period
  Interventions: Device: Sham Device

INTERVENTIONS:
Device: Wrist Device — peripheral nerve stimulation via wrist-worn device
  Arms: Wrist Device
Device: Ear Device — peripheral nerve stimulation via ear-worn device
  Arms: Ear Device
Device: Sham Device — Wrist-worn device that does not actually deliver stimulation
  Arms: Sham Device

SUMMARY:
This is a three-arm, single-blinded, randomized, sham-controlled, nonsignificant risk study to assess the feasibility of reducing Atrial Fibrillation burden with peripheral nerve stimulation. The three arms include treatment with a wrist-worn neuromodulation ("wrist device"), treatment with an ear-worn neuromodulation device ("ear device") and sham stimulation with wrist-worn device that does not actually deliver stimulation ("sham device"). ECG patches will be worn on the chest to measure AF episode onset and duration ("ECG Patch"). Additionally, a wrist-worn monitoring device will be used for the measurement of heart rate (HR), heart rate variability (HRV), and other biomarkers ("Cardiac Measurement Device (CMD)"). Finally, subjects will track AF episode onset, duration, and symptom type in an AF diary.

ELIGIBILITY:
Inclusion Criteria:

* At least 22 years of age and less than 80 years of age
* Diagnosed with paroxysmal atrial fibrillation, as documented on ECG, trans-telephonic monitoring (TTM), cardiac event monitoring, Holter monitoring, or implantable loop recording (episodes must be longer than 30 seconds to qualify)
* At least one symptomatic atrial fibrillation episodes per month over the last three months
* AF burden of at least 5%, as measured within the past 3 months, with no change in AF treatment since measurement
* Willing to stay on stable medications for the duration of the study
* Able and willing to use their smartphone to download the application associated with the Cardiac Measurement Device
* Competent and willing to provide written, informed consent to participate in the study

Exclusion Criteria:

* Prior cardiac ablation, or cardiac ablation planned within 6 weeks of Visit 1
* Cardioversion procedure performed within the last 12 weeks
* Valvular atrial fibrillation by transthoracic echocardiography
* Left atrial anteroposterior diameter greater than 5.5 cm by transthoracic echocardiography
* Prior or planned cardiac transplantation or cardiac surgery
* Cerebral ischemic event (stroke or transient ischemic attack) within the last 6 months
* Myocardial infarction within the last 6 months
* Heart failure (NYHA class III or IV)
* Left ventricular ejection fraction less than 35%
* Recurrent vaso-vagal syncopal episodes
* Unilateral or bilateral vagotomy
* Hemodynamic instability
* Structural heart damage
* Implanted active electrical medical device, such as pacemaker, implantable loop recorders, defibrillator, or deep brain stimulator
* Implanted metal or electrical devices in the head or treated hand
* Not currently on anticoagulants
* History of epilepsy or seizures
* Peripheral neuropathy affecting the upper left extremity
* Pregnancy, anticipated pregnancy, or nursing during the study
* Unable or unwilling to comply fully with study procedures and followup, including atrial fibrillation diary requirements
* Known allergy to any of the device materials that are in contact with prospective subject's skin
* Current participation, or previous participation within the last 30 days, in another interventional clinical trial that may confound the results of this study, unless otherwise approved by the Sponsor
* Subjects unable to communicate with the Investigator and study staff
* Presence of any health condition that should preclude participation in this study, per the Investigator's opinion

Ages: 22 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of time spent in AF during the 4-week treatment period compared to the 2-week run-in period (prior to treatment) for AF episodes >= 30 seconds duration | 6 weeks

SECONDARY OUTCOMES:
Time to first recurrence of any AF (>= 30 seconds duration) during treatment period compared to run-in period | 6 weeks
Time to first recurrence of symptomatic AF during treatment period compared to run-in period | 6 weeks
Average AF episode duration during the treatment period compared to the run-in period (for episodes >= 30seconds duration) | 6 weeks
Number of AF episodes lasting >= 5.5 hours | 6 weeks
Average duration of ongoing AF episodes (>= 30 seconds duration) following the start of therapy sessions | 6 weeks
Atrial Fibrillation Effect on Quality of Life (AFEQL) score at the end of the treatment period compared to end of the run-in period | 6 weeks
Compliance to per-protocol therapy measured by the percentage of full and partial therapy sessions delivered relative to total sessions required per-protocol | 6 weeks
Compliance of daily therapy measured by the percentage of treatment days subjects performed full or partial therapy sessions | 6 weeks

OTHER OUTCOMES:
Number of AF-related emergency visits | 6 weeks
Number of AF-related in-patient hospitalizations | 6 weeks
Number of cardioversion procedures | 6 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Mayo Clinic, Rochester, Minnesota
  - Medical University of South Carolina, Charleston, South Carolina